CLINICAL TRIAL: NCT02900911
Title: Effects of Prophylactic Swallowing Exercises on Dysphagia and Quality of Life in Patients With Head and Neck Cancer Receiving Radiotherapy: A Randomized Clinical Trial
Brief Title: Swallowing Rehabilitation in Patients With Head and Neck Cancer Receiving Radiotherapy
Acronym: ReDyOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Collaborators: Asociación Española contra el Cáncer (Other)
Responsible Party: Principal Investigator, Esther Marco Navarro, PhD, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2014/5707/l
Record Dates: First submitted 2016-02-15; First posted 2016-09-14 (Estimated); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Cancer of Head and Neck
Keywords: head and neck cancer; dysphagia; rehabilitation; radiation therapy
MeSH Terms: conditions — Head and Neck Neoplasms; Deglutition Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early rehabilitation (Experimental): Early intervention consisting in standard swallow therapy and instructions to train respiratory muscles starting 2 weeks before Radiotherapy during 6 months
  Interventions: Other: Early rehabilitation
- Later rehabilitation (Active Comparator): Late intervention consists of standard swallow therapy and instructions to train respiratory muscles starting after completing Radiotherapy
  Interventions: Other: Late rehabilitation

INTERVENTIONS:
Other: Early rehabilitation — Early swallowing exercises and respiratory muscle training: Standard swallow therapy and instructions for training submental muscles involved in swallowing function and expiratory strength starting 2 weeks before radiotherapy
  Expiratory/Inspiratory training: the training load is the maximum inspiratory/expiratory load defined according to patient tolerance. This load will be equivalent to 10 maximal repetitions (RM) as 10 consecutive inspirations (x 5 sessions), three times a day.
  All sessions will be conducted under the supervision of an expert physiotherapist/swallowing therapist. The total duration of the training program is 6 months.
  Arms: Early rehabilitation
Other: Late rehabilitation — Late swallowing exercises and respiratory muscle training: Standard swallow therapy and instructions for training submental muscles involved in swallowing function and expiratory strength starting after completing radiotherapy
  Arms: Later rehabilitation

SUMMARY:
Head and neck cancer has a negative impact in swallowing function and quality of life. Rehabilitation has proven its usefulness after radiation therapy (RT), but some studies suggest that interventions should be initiated prior to RT sessions. This study aims to evaluate the effects of prophylactic rehabilitation on swallowing and quality of life. The study pretends to establish a preventive rehabilitative program with the target of reducing RT side effects and improve patients' quality of life.

DETAILED DESCRIPTION:
Head and neck cancer has a negative impact in swallowing function and quality of life. Although current diagnostic and therapeutic protocols try to preserve swallowing and speaking, acute or late dysphagia as well as a poor quality of life are frequent in these patients.

Some studies have reported an improvement in swallowing function after an exercise based intervention following radiation therapy (RT), regardless the need of concomitant chemotherapy (RT-QT). Other studies focus the interest in the use of prophylactic exercises to prevent or minimize post-swallowing dysfunction.

Patients receiving RT or RT-QT refer worsening of their quality of life, especially during the first days after treatment. One study suggests that rehabilitation prior to cancer treatment could potentially improve quality of life. However, this observation should be contrasted with a randomized study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced head and neck cancer receiving radiotherapy

Exclusion Criteria:

* Candidates to surgical treatment
* Previous head and neck cancer
* Dysphagia due to causes other than cancer
* Previous head or neck radiation therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-05; Primary Completion 2020-04 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Change in dysphagia severity at three months post radiotherapy | 2 weeks before beginning radiotherapy, and 3 months after completing radiotherapy
  8-point Penetration Aspiration Scale: scores of 1-2 indicate normal swallowing, 3-5 reflect penetration, and >6, aspiration
Change in quality of life at three months post radiotherapy | 2 weeks before beginning radiotherapy and 3 months after completing radiotherapy
  Head & Neck Cancer 35 (HN35)

SECONDARY OUTCOMES:
Change in dysphagia security signs at three months post radiotherapy | 2 weeks before beginning radiotherapy and 3 months after completing radiotherapy
  Security signs (tone of voice, coughing during or after eating, or desaturation of more than 3% compared to baseline pulse oximetry) assessed with the Volume Viscosity Swallow Test
Change in lingual Force at three months post radiotherapy | 2 weeks before beginning radiotherapy and 3 months after completing radiotherapy
  Lingual Force: maximum isometric tongue pressure of three peak isometric tongue pressure scores assessed with the IOPI system.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de l'Esperança, Barcelona, Spain

REFERENCES:
- [Background] Stenson KM, MacCracken E, List M, Haraf DJ, Brockstein B, Weichselbaum R, Vokes EE. Swallowing function in patients with head and neck cancer prior to treatment. Arch Otolaryngol Head Neck Surg. 2000 Mar;126(3):371-7. doi: 10.1001/archotol.126.3.371. PMID 10722011
- [Background] Quer M, Leon X, Orus C, Recher K, Gras JR. [Analysis of 2,500 squamous cell carcinoma of the head and neck]. Acta Otorrinolaringol Esp. 2001 Apr;52(3):201-5. doi: 10.1016/s0001-6519(01)78198-8. Spanish. PMID 11526864
- [Background] Kulbersh BD, Rosenthal EL, McGrew BM, Duncan RD, McColloch NL, Carroll WR, Magnuson JS. Pretreatment, preoperative swallowing exercises may improve dysphagia quality of life. Laryngoscope. 2006 Jun;116(6):883-6. doi: 10.1097/01.mlg.0000217278.96901.fc. PMID 16735913
- [Background] Carroll WR, Locher JL, Canon CL, Bohannon IA, McColloch NL, Magnuson JS. Pretreatment swallowing exercises improve swallow function after chemoradiation. Laryngoscope. 2008 Jan;118(1):39-43. doi: 10.1097/MLG.0b013e31815659b0. PMID 17989581
- [Background] Lazarus CL. Effects of chemoradiotherapy on voice and swallowing. Curr Opin Otolaryngol Head Neck Surg. 2009 Jun;17(3):172-8. doi: 10.1097/MOO.0b013e32832af12f. PMID 19337126
- [Background] Dirix P, Abbeel S, Vanstraelen B, Hermans R, Nuyts S. Dysphagia after chemoradiotherapy for head-and-neck squamous cell carcinoma: dose-effect relationships for the swallowing structures. Int J Radiat Oncol Biol Phys. 2009 Oct 1;75(2):385-92. doi: 10.1016/j.ijrobp.2008.11.041. Epub 2009 Jun 24. PMID 19553033
- [Background] Murphy BA, Gilbert J. Dysphagia in head and neck cancer patients treated with radiation: assessment, sequelae, and rehabilitation. Semin Radiat Oncol. 2009 Jan;19(1):35-42. doi: 10.1016/j.semradonc.2008.09.007. PMID 19028344
- [Background] Platteaux N, Dirix P, Dejaeger E, Nuyts S. Dysphagia in head and neck cancer patients treated with chemoradiotherapy. Dysphagia. 2010 Jun;25(2):139-52. doi: 10.1007/s00455-009-9247-7. Epub 2009 Aug 27. PMID 19711127
- [Background] Tang Y, Shen Q, Wang Y, Lu K, Wang Y, Peng Y. A randomized prospective study of rehabilitation therapy in the treatment of radiation-induced dysphagia and trismus. Strahlenther Onkol. 2011 Jan;187(1):39-44. doi: 10.1007/s00066-010-2151-0. Epub 2010 Dec 10. PMID 21136031
- [Background] Roe JW, Ashforth KM. Prophylactic swallowing exercises for patients receiving radiotherapy for head and neck cancer. Curr Opin Otolaryngol Head Neck Surg. 2011 Jun;19(3):144-9. doi: 10.1097/MOO.0b013e3283457616. PMID 21430531
- [Background] Lin PH, Hsiao TY, Chang YC, Ting LL, Chen WS, Chen SC, Wang TG. Effects of functional electrical stimulation on dysphagia caused by radiation therapy in patients with nasopharyngeal carcinoma. Support Care Cancer. 2011 Jan;19(1):91-9. doi: 10.1007/s00520-009-0792-2. Epub 2009 Nov 29. PMID 20091057
- [Background] Kotz T, Federman AD, Kao J, Milman L, Packer S, Lopez-Prieto C, Forsythe K, Genden EM. Prophylactic swallowing exercises in patients with head and neck cancer undergoing chemoradiation: a randomized trial. Arch Otolaryngol Head Neck Surg. 2012 Apr;138(4):376-82. doi: 10.1001/archoto.2012.187. PMID 22508621
- [Background] Tedla M, Valach M, Carrau RL, Varga I, Profant M, Mraz P, Weismann P. Impact of radiotherapy on laryngeal intrinsic muscles. Eur Arch Otorhinolaryngol. 2012 Mar;269(3):953-8. doi: 10.1007/s00405-011-1686-8. Epub 2011 Jul 8. PMID 21739096
- [Background] Russi EG, Corvo R, Merlotti A, Alterio D, Franco P, Pergolizzi S, De Sanctis V, Ruo Redda MG, Ricardi U, Paiar F, Bonomo P, Merlano MC, Zurlo V, Chiesa F, Sanguineti G, Bernier J. Swallowing dysfunction in head and neck cancer patients treated by radiotherapy: review and recommendations of the supportive task group of the Italian Association of Radiation Oncology. Cancer Treat Rev. 2012 Dec;38(8):1033-49. doi: 10.1016/j.ctrv.2012.04.002. Epub 2012 Apr 27. PMID 22542950
- [Background] Hutcheson KA, Lewin JS, Barringer DA, Lisec A, Gunn GB, Moore MW, Holsinger FC. Late dysphagia after radiotherapy-based treatment of head and neck cancer. Cancer. 2012 Dec 1;118(23):5793-9. doi: 10.1002/cncr.27631. Epub 2012 May 17. PMID 23640737
- [Background] Wall LR, Ward EC, Cartmill B, Hill AJ. Physiological changes to the swallowing mechanism following (chemo)radiotherapy for head and neck cancer: a systematic review. Dysphagia. 2013 Dec;28(4):481-493. doi: 10.1007/s00455-013-9491-8. PMID 24078216
- [Background] Citak E, Tulek Z. Longitudinal quality of life in Turkish patients with head and neck cancer undergoing radiotherapy. Support Care Cancer. 2013 Aug;21(8):2171-83. doi: 10.1007/s00520-013-1774-y. Epub 2013 Mar 9. PMID 23475195
- [Background] Long YB, Wu XP. A randomized controlled trail of combination therapy of neuromuscular electrical stimulation and balloon dilatation in the treatment of radiation-induced dysphagia in nasopharyngeal carcinoma patients. Disabil Rehabil. 2013 Mar;35(6):450-4. doi: 10.3109/09638288.2012.697250. Epub 2012 Jul 4. PMID 22762238
- [Background] Rathod S, Gupta T, Ghosh-Laskar S, Murthy V, Budrukkar A, Agarwal J. Quality-of-life (QOL) outcomes in patients with head and neck squamous cell carcinoma (HNSCC) treated with intensity-modulated radiation therapy (IMRT) compared to three-dimensional conformal radiotherapy (3D-CRT): evidence from a prospective randomized study. Oral Oncol. 2013 Jun;49(6):634-42. doi: 10.1016/j.oraloncology.2013.02.013. Epub 2013 Apr 4. PMID 23562564